CLINICAL TRIAL: NCT04345744
Title: Evaluation of the Rinse With Chlorhexidine Plus Hyaluronic Acid Mouthwash in Periodontal Surgical Wound Healing
Acronym: CLOR_3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Full Professor of Periodontology, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CLOR_3
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Periodontal Diseases; Periodontal Pocket
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket

STUDY DESIGN:
Intervention Model Description: Single-centre randomized, parallel design, clinical trial with a 2 week follow-up
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After surgery, patients will be randomly assigned to study groups corresponding to mouth rinse prescription. The mouth rinse will be assigned by an experimenter not involved in the following steps of the study, in order to maintain the examiner blind. The patient will receive a non-labelled mouth rinse to avoid biases both of the examiner and the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1 (Experimental): administration of a hyaluronic and 0.2% chlorhexidine mouth rinse
  Interventions: Procedure: Periodontal surgery; Device: Hyaluronic and 0.2% chlorhexidine mouth rinse
- Test group 2 (Experimental): administration of chlorhexidine 0.2% mouth rinse
  Interventions: Procedure: Periodontal surgery; Device: Chlorhexidine 0.2% mouth rinse
- Control Group (Active Comparator): No administration of mouth rinses after surgery
  Interventions: Procedure: Periodontal surgery

INTERVENTIONS:
Procedure: Periodontal surgery — Surgery will be performed following a standardized protocol by a single operator (FG). The procedure consists in the performance of a primary full-thickness flap incision, and of a secondary releasing vertical incision of maximum 3 mm limited to keratinized gingiva. At the end of the surgical procedure, soft tissues will be repositioned by means of a suture involving only the primary incision, while it will not be performed on the releasing incision.
Device: Hyaluronic and 0.2% chlorhexidine mouth rinse — The mouth rinse protocol assigned to each study participant included a 10 ml-rinse for 60 seconds twice-a-day (every 12 hours) for 14 days.
  Arms: Test group 1
Device: Chlorhexidine 0.2% mouth rinse — The mouth rinse protocol assigned to each study participant included a 10 ml-rinse for 60 seconds twice-a-day (every 12 hours) for 14 days.
  Arms: Test group 2

SUMMARY:
Evaluate the response of the gingival tissues to the use of mouthwash with chlorhexidine and chlorhexidine + hyaluronic acid in terms of healing of the periodontal surgical wound.

DETAILED DESCRIPTION:
Patients included in the study will undergo a thorough clinical examination aiming at collecting all the data desired: periodontal parameters of Probing Pocket Depth (PPD) and presence of recession of the gingival margin (Rec) will be recorded on six sites/tooth in the area selected for periodontal surgery by a single calibrated examiner using a University of North Carolina (UNC) 15-mm periodontal probe at a 0.3 N probing pressure. Surgery will be performed following a standardized protocol by a single operator.

After surgery, patients will be randomly assigned to study groups corresponding to mouth rinse prescription. The mouth rinse will be assigned by an experimenter not involved in the following steps of the study, in order to maintain the examiner blind. The patient will receive a non-labelled mouth rinse to avoid biases both of the examiner and the patient. The patient will also be given a diary for the registration of the number of rinses per day, to be returned to the examiner at T14. The mouth rinse protocol assigned to each study participant includes a 10 ml-rinse for 60 seconds twice-a-day (every 12 hours) for 14 days.

The patients will be allocated in one of the three distinct study groups as it follows:

* Group A: no administration of mouth rinses after surgery (control group)
* Group B: administration of a hyaluronic and 0.2% chlorhexidine mouth rinse (test group 1)
* Group C: administration of chlorhexidine 0.2% mouth rinse (test group 2).

Post-treatment photographs of surgical incision will be taken immediately after periodontal surgery and at 3 (T3), 7 (T7), and 14 (T14) days post-op, in order to allow the evaluation of the degree of wound healing. The degree of surgical healing will be evaluated using the Periodontal Wound Healing Index (Wachtel classification) on all the incisions, and a score from 1 to 5 will be assigned.

At T3, T7, and T14 the following clinical parameters will be recorded for each tooth in the surgical area: PPD, Rec, PI, and BOP. The clinical examinations will be performed by calibrated examiner blind to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* males or females of age range between 18 and 70 years,
* good health status,
* indication to perform periodontal surgery,
* patients willing to give informed consent,
* compliance to the study follow-up,
* plaque index (PI) score 0 and
* bleeding on probing (BOP) <25%

Exclusion Criteria:

* pregnancy or breast-feeding,
* therapy with oral contraceptives,
* indication to antibiotic therapy prior to surgical treatment,
* chronic infections,
* systemic diseases (including cardiovascular, pulmonary, cerebral, and metabolic diseases),
* previous therapy with the mouth rinses employed in the present study, and
* smoking habit (>20 cigarettes per day, and/or pipe or cigar smoking).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth (PPD) | Measured at Baseline and at day 3, day 7, and day 14
  Changes in PPD, measured orally through clinical examination. Unit of measure: mm

SECONDARY OUTCOMES:
Clinical attachment level (CAL) | Measured at Baseline and at day 3, day 7, and day 14
  Changes in CAL , measured orally through clinical examination. Unit of measure: mm
Recession of the gingival margin (REC) | Measured at Baseline and at day 3, day 7, and day 14
  Changes in REC, measured orally through clinical examination. Unit of measure: mm
Bleeding on probing (BOP) | Measured at Baseline
  BOP, measured orally through clinical examination. Unit of measure: %
Angulated bleeding index (AngBI) | Measured at day 3, day 7, and day 14
  AngBI, measured orally through clinical examination. Unit of measure: %
Plaque index (PI) | Measured at Baseline and at day 3, day 7, and day 14
  Changes in PI, measured orally through clinical examination. Unit of measure: %
Periodontal Wound Healing Index (PWHI) (Wachtel classification) | Measured at day 3, day 7, and day 14
  Changes in PWHI, measured orally through clinical examination on all the incisions, assigning a score from 1 to 5.
  * Score 1: complete wound healing: absence of fibrin line in the interproximal area
  * Score 2: complete wound healing: presence of a thin fibrin line in the interproximal area
  * Score 3: complete wound healing: presence of fibrin clot in the interproximal area
  * Score 4: incomplete wound healing: presence of partial necrosis of the interproximal area
  * Score 5: incomplete wound healing: total necrosis of the interproximal area
Post-surgical photographs | Taken at Baseline, day 3, day 7, and day 14
  Post-surgical photographs will be taken and analysed after the completion of the trial

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berchier CE, Slot DE, Van der Weijden GA. The efficacy of 0.12% chlorhexidine mouthrinse compared with 0.2% on plaque accumulation and periodontal parameters: a systematic review. J Clin Periodontol. 2010 Sep;37(9):829-39. doi: 10.1111/j.1600-051X.2010.01575.x. Epub 2010 Jul 7. PMID 20618550